CLINICAL TRIAL: NCT01015911
Title: A Phase 1, Open-label, Dose-escalation Study to Evaluate the Safety and Tolerability of SGN-75 in Patients With CD70-positive Relapsed or Refractory Non-Hodgkin Lymphoma or Metastatic Renal Cell Carcinoma
Brief Title: A Phase 1 Dose-escalation Trial of SGN-75 in CD70-positive Non-Hodgkin Lymphoma or Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN75-001
Record Dates: First submitted 2009-11-13; First posted 2009-11-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Carcinoma, Renal Cell; Lymphoma, Non-Hodgkin
Keywords: Antibodies, Monoclonal; Antibody-Drug Conjugate; Antigens, CD70; Lymphoma, Non-Hodgkin; Carcinoma, Renal Cell; Immunotherapy; Drug Therapy; monomethylauristatin F
MeSH Terms: conditions — Carcinoma, Renal Cell; Lymphoma, Non-Hodgkin | interventions — SGN-75 antibody-drug conjugate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): SGN-75
  Interventions: Drug: SGN-75

INTERVENTIONS:
Drug: SGN-75 — SGN-75 (IV) in 21- or 28-day cycles; dose range: 0.3-9 mg/kg

SUMMARY:
This is a phase 1, open-label, dose-escalation clinical trial to evaluate the safety of SGN-75 in patients with CD70-positive relapsed or refractory non-Hodgkin lymphoma or metastatic renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-confirmed diagnosis of NHL or RCC
* Relapsed, refractory, or progressive disease following at least 1 prior systemic therapy
* Confirmed CD70 expression
* Measurable disease, defined as at least 1 lesion >1.5 cm in the greatest transverse diameter for patients with NHL, and at least 1 non-resectable tumor lesion > or equal to 10 mm in diameter for patients with RCC

Exclusion Criteria:

* Previously received an allogeneic transplant
* History of another primary malignancy that has not been in remission for at least 3 years
* Prior anti-CD70-directed therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and laboratory abnormalities | Through 1 month following last dose

SECONDARY OUTCOMES:
Best clinical response | Every 2 months
Duration of response, progression-free survival | Every 3 months until progression of disease or initiation of new treatment for cancer
Blood concentrations of SGN-75 and metabolites | Through 1 month following last dose
Incidence of antitherapeutic antibodies | Through 1 month following last dose

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Whiting, PharmD, BCOP, Study Director — Seagen Inc.
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - UCLA Medical Center / University of California at Los Angeles, Los Angeles, California
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Seattle Cancer Care Alliance / University of Washington, Seattle, Washington

REFERENCES:
- [Result] Tannir NM, Forero-Torres A, Ramchandren R, Pal SK, Ansell SM, Infante JR, de Vos S, Hamlin PA, Kim SK, Whiting NC, Gartner EM, Zhao B, Thompson JA. Phase I dose-escalation study of SGN-75 in patients with CD70-positive relapsed/refractory non-Hodgkin lymphoma or metastatic renal cell carcinoma. Invest New Drugs. 2014 Dec;32(6):1246-57. doi: 10.1007/s10637-014-0151-0. Epub 2014 Aug 22. PMID 25142258